CLINICAL TRIAL: NCT07047755
Title: Trastuzumab Rezetecan Plus Pertuzumab as Neoadjuvant Treatment for Early or Locally Advanced HER2-positive Breast Cancer：A Prospective, Open-label, Phase II Trial
Brief Title: Trastuzumab Rezetecan Plus Pertuzumab in the Neoadjuvant Treatment of HER2 Positive BC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-027
Record Dates: First submitted 2025-06-19; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Trastuzumab Rezetecan; Pertuzumab
  Interventions: Drug: Trastuzumab Rezetecan; Drug: Pertuzumab

INTERVENTIONS:
Drug: Trastuzumab Rezetecan — Trastuzumab Rezetecan
Drug: Pertuzumab — Pertuzumab

SUMMARY:
This is a prospective, open-label, phase II study evaluating the efficacy and safety of Trastuzumab Rezetecan in combination with pertuzumab in early or locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
Patients with early-stage or locally advanced HER2-positive breast cancer were planned to be enrolled and subjected to neoadjuvant therapy with the regimen of Trastuzumab Rezetecan combined with Pertuzumab. The primary objective was to evaluate the efficacy and safety of Trastuzumab Rezetecan plus Pertuzumab as neoadjuvant treatment for early-stage or locally advanced HER2-positive breast cancer. Subjects will continue medication until surgery is completed, or until disease progression, intolerable toxicity, withdrawal of informed consent, or when the investigator determines that medication must be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years;
2. Histopathologically confirmed HER2 positive breast cancer;
3. Patients were diagnosed with stage II-III breast cancer;
4. At least one measurable target lesion according to RECIST V1.1;
5. ECOG performance status score of 0 to 1;
6. Life expectancy ≥12 weeks;
7. Adequate bone marrow reserve and organ system function reserve;
8. Participants should be able and willing to comply with the study protocol requirement;

Exclusion Criteria:

1. Breast cancer not histologically confirmed;
2. Known inherited or acquired bleeding and thrombotic tendencies;
3. Known allergy or contraindication to the study drug and its excipients;
4. Previously been treated with any anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
5. Concurrent receipt of any other form of anti-cancer therapy;
6. History of a second primary malignancy, except for adequately treated skin cancer;
7. Participation in other drug clinical trials within 4 weeks before enrollment;
8. Major surgical procedures unrelated to breast cancer within 4 weeks prior to the first drug administration, or not fully recovered from such procedures;
9. Presence of any active autoimmune disease or history of autoimmune disease with potential for recurrence;
10. Uncontrolled or significant cardiovascular and cerebrovascular diseases;
11. Subjects with known or suspected interstitial pneumonia;
12. Presence of active hepatitis B, hepatitis C, liver cirrhosis;
13. Pregnant or lactating female patients;
14. History of definite neurological or mental disorders, or any other conditions that the investigator believes make the patient unsuitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
pCR rate | At the time of surgery
  Total pathological complete response (tpCR: ypT0-is，ypN0)

SECONDARY OUTCOMES:
iDFS | Up to approximately 5 years
  Invasive disease-free survival
EFS | Up to approximately 5 years
  Event-free survival
ORR | Up to approximately 24 weeks after the first administration
  Objective Response Rate
AEs | From the first dose until 30 days after last dose
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) according to CTCAE 5.0